CLINICAL TRIAL: NCT01376271
Title: Special Drug Use Investigation for PAXIL (Paroxetine) Social Anxiety Disorder (Long-term)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114102
Record Dates: First submitted 2011-06-09; First posted 2011-06-20 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Social Phobia
MeSH Terms: conditions — Phobia, Social | interventions — Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects prescribed paroxetine tablets: Subjects with SAD prescribed paroxetine tablets during study period
  Interventions: Drug: Paroxetine

INTERVENTIONS:
Drug: Paroxetine

SUMMARY:
The study is designed to evaluate the safety and efficacy of paroxetine on the long-term use in Japanese Social Anxiety Disorder (SAD) subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are diagnosed as having SAD
* Subjects who are expected to use paroxetine tablets for the first time

Exclusion Criteria:

* Subjects taking pimozide
* Subjects taking monoamine oxidase (MAO) inhibitor or within two weeks after discontinuation of MAO inhibitor
* Subjects with hypersensitivity to paroxetine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects diagnosed as having social anxiety disorder (SAD) are to be given paroxetine tablets according to the prescribing information
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2010-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The number of adverse events in Japanese subjects with social anxiety disorder treated with paroxetine tablets | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline